CLINICAL TRIAL: NCT00005686
Title: Dietary Intervention Methods for Clinical Trials
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4171; R01HL041332 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To develop a dietary intervention method that was capable of producing large sustained weight losses and was thus suitable for use in clinical trials related to obesity.

DETAILED DESCRIPTION:
BACKGROUND:

A study by the investigators showed that a method based on principles of antecedent control, namely the provision of food to participants, was successful in almost doubling weight losses over a twelve month period compared to those attained in a standard behavioral weight control program. These weight losses were associated with substantial improvements in cardiovascular risk factors.

DESIGN NARRATIVE:

There were several studies in this two-center project (R01HL41330 and R01HL41332). Obese subjects, male and female, were recruited at the University of Pittsburgh and the University of Minnesota. The subjects were randomly assigned to one of five treatment groups: no treatment control, standard behavioral nutrition program, standard program with incentives, standard program with food provision, and standard program with both incentives and food provision. The effectiveness of the treatments was analyzed by assessing changes in body weight, coronary heart disease risk factors (lipids, blood pressure, insulin, and glucose) and process variables (eating and exercise behavior, knowledge, barriers to adherence) at six month intervals for eighteen months.

The project was renewed in April 1992 and included four studies. Study 1 determined whether there were long-term benefits to food provision by reexamining the 202 participants in the original study one year after the end of treatment. Study 2 investigated the factors related to the successful food provision intervention by comparing the additive effects of standard behavioral treatment and the three central components of food provision: structured meal plans, prepackaged food and subsidy of the food. It also explored theoretical mechanisms which might underlie the food provision effect, specifically decision making and stimulus control. Study 3 evaluated the effectiveness of extending the food provision methodology to families. Overweight spouse pairs were randomized to treatments in which either one member of the pair participated in treatment and received food, or both members of the pair participated and were provided with food. Study 4 determined whether the principles of antecedent control could also be applied to exercise. Participants were randomized to weight control programs which included either the usual exercise instructions or structured plans for exercise and free passes to exercise facilities near their home. It was hypothesized that providing food for the obese spouse as well as the patient, and providing antecedent control for exercise through structured plans and free passes would both improve the maintenance of weight loss.

The studies were renewed in FY 1998 through April, 2002 to compare the long-term weight losses achieved in a standard behavioral program with those obtained in an enhanced exercise intervention. The exercise goal in the standard program was 1000 kcal/week, while that in the enhanced exercise program was 2500 kcal/week. The study was conducted with 180 subjects divided equally between men and women, half recruited in Minneapolis and the other half in Pittsburgh. The primary hypotheses were that the enhanced exercise intervention group would have significantly greater weight losses than the standard intervention group at the end of the 18 month treatment program and at the 30-month follow-up. In addition, the two conditions were compared at 0, 6, 12, 18, and 30 months with regard to exercise levels, variables that might be related to exercise and weight loss, and measures related to quality of life. Furthermore, the investigators attempted to determine predictors of long-term weight loss and exercise behavior, and examined the effects of social support on exercise level and weight loss of the enhanced exercise intervention group.

Include both R01HL41330 and R01HL41332.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-04; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jeffery — University of Minnesota; Rena Wing — The Miriam Hospital

REFERENCES:
- [Background] Wing RR. Physical activity in the treatment of the adulthood overweight and obesity: current evidence and research issues. Med Sci Sports Exerc. 1999 Nov;31(11 Suppl):S547-52. doi: 10.1097/00005768-199911001-00010. PMID 10593526
- [Background] Wing RR, Jeffery RW. Benefits of recruiting participants with friends and increasing social support for weight loss and maintenance. J Consult Clin Psychol. 1999 Feb;67(1):132-8. doi: 10.1037//0022-006x.67.1.132. PMID 10028217
- [Background] Jeffery RW, Wing RR, Thorson C, Burton LR. Use of personal trainers and financial incentives to increase exercise in a behavioral weight-loss program. J Consult Clin Psychol. 1998 Oct;66(5):777-83. doi: 10.1037//0022-006x.66.5.777. PMID 9803696
- [Background] Jeffery RW, Wing RR, Mayer RR. Are smaller weight losses or more achievable weight loss goals better in the long term for obese patients? J Consult Clin Psychol. 1998 Aug;66(4):641-5. doi: 10.1037//0022-006x.66.4.641. PMID 9735580
- [Background] Wirfalt AK, Jeffery RW. Using cluster analysis to examine dietary patterns: nutrient intakes, gender, and weight status differ across food pattern clusters. J Am Diet Assoc. 1997 Mar;97(3):272-9. doi: 10.1016/s0002-8223(97)00071-0. PMID 9060944
- [Background] Wing RR. Insulin sensitivity as a predictor of weight regain. Obes Res. 1997 Jan;5(1):24-9. doi: 10.1002/j.1550-8528.1997.tb00279.x. PMID 9061712
- [Background] Wing RR, Sinha MK, Considine RV, Lang W, Caro JF. Relationship between weight loss maintenance and changes in serum leptin levels. Horm Metab Res. 1996 Dec;28(12):698-703. doi: 10.1055/s-2007-979881. PMID 9013745
- [Background] Wing RR, Jeffery RW, Pronk N, Hellerstedt WL. Effects of a personal trainer and financial incentives on exercise adherence in overweight women in a behavioral weight loss program. Obes Res. 1996 Sep;4(5):457-62. doi: 10.1002/j.1550-8528.1996.tb00254.x. PMID 8885210
- [Background] Jeffery RW, Wing RR. Long-term effects of interventions for weight loss using food provision and monetary incentives. J Consult Clin Psychol. 1995 Oct;63(5):793-6. doi: 10.1037//0022-006x.63.5.793. PMID 7593872
- [Background] Wing RR. Changing diet and exercise behaviors in individuals at risk for weight gain. Obes Res. 1995 Sep;3 Suppl 2:277s-282s. doi: 10.1002/j.1550-8528.1995.tb00474.x. PMID 8581787
- [Background] Wing RR, Jeffery RW, Hellerstedt WL. A prospective study of effects of weight cycling on cardiovascular risk factors. Arch Intern Med. 1995 Jul 10;155(13):1416-22. PMID 7794091
- [Background] Wing RR, Jeffery RW. Effect of modest weight loss on changes in cardiovascular risk factors: are there differences between men and women or between weight loss and maintenance? Int J Obes Relat Metab Disord. 1995 Jan;19(1):67-73. PMID 7719395
- [Background] French SA, Jeffery RW, Wing RR. Sex differences among participants in a weight-control program. Addict Behav. 1994 Mar-Apr;19(2):147-58. doi: 10.1016/0306-4603(94)90039-6. PMID 8036962
- [Background] Jeffery RW, Wing RR, Thorson C, Burton LR, Raether C, Harvey J, Mullen M. Strengthening behavioral interventions for weight loss: a randomized trial of food provision and monetary incentives. J Consult Clin Psychol. 1993 Dec;61(6):1038-45. doi: 10.1037//0022-006x.61.6.1038. PMID 8113481
- [Background] Bunker CH, Wing RR, Becker DJ, Kuller LH. Sodium-lithium countertransport activity is decreased after weight loss in healthy obese men. Metabolism. 1993 Aug;42(8):1052-8. doi: 10.1016/0026-0495(93)90022-g. PMID 8345810
- [Background] Wing RR, Jeffery RW, Burton LR, Thorson C, Kuller LH, Folsom AR. Change in waist-hip ratio with weight loss and its association with change in cardiovascular risk factors. Am J Clin Nutr. 1992 Jun;55(6):1086-92. doi: 10.1093/ajcn/55.6.1086. PMID 1595579
- [Background] Wing RR. Behavioral treatment of severe obesity. Am J Clin Nutr. 1992 Feb;55(2 Suppl):545S-551S. doi: 10.1093/ajcn/55.2.545s. PMID 1733124
- [Background] Wing RR. Obesity and weight gain during adulthood: a health problem for United States women. Womens Health Issues. 1992 Summer;2(2):114-20; discussion 120-2. doi: 10.1016/s1049-3867(05)80279-8. No abstract available. PMID 1617307
- [Background] Hellerstedt WL, Jeffery RW. The effects of a telephone-based intervention on weight loss. Am J Health Promot. 1997 Jan-Feb;11(3):177-82. doi: 10.4278/0890-1171-11.3.177. PMID 10165095
- [Background] Hennrikus DJ, Jeffery RW. Worksite intervention for weight control: a review of the literature. Am J Health Promot. 1996 Jul-Aug;10(6):471-98. doi: 10.4278/0890-1171-10.6.471. PMID 10163312
- [Background] Jeffery RW, French SA, Raether C, Baxter JE. An environmental intervention to increase fruit and salad purchases in a cafeteria. Prev Med. 1994 Nov;23(6):788-92. doi: 10.1006/pmed.1994.1135. PMID 7855111
- [Background] Jeffery RW, Drewnowski A, Epstein LH, Stunkard AJ, Wilson GT, Wing RR, Hill DR. Long-term maintenance of weight loss: current status. Health Psychol. 2000 Jan;19(1S):5-16. doi: 10.1037/0278-6133.19.suppl1.5. PMID 10709944
- [Background] Wing RR, Jeffery RW. Food provision as a strategy to promote weight loss. Obes Res. 2001 Nov;9 Suppl 4:271S-275S. doi: 10.1038/oby.2001.130. PMID 11707553
- [Background] Wing RR, Hill JO. Successful weight loss maintenance. Annu Rev Nutr. 2001;21:323-41. doi: 10.1146/annurev.nutr.21.1.323. PMID 11375440
- [Background] Wing RR. Behavioral interventions for obesity: recognizing our progress and future challenges. Obes Res. 2003 Oct;11 Suppl:3S-6S. doi: 10.1038/oby.2003.219. No abstract available. PMID 14569033
- [Background] Wing RR, Gorin AA. Behavioral techniques for treating the obese patient. Prim Care. 2003 Jun;30(2):375-91. doi: 10.1016/s0095-4543(03)00009-5. PMID 14567154
- [Background] Jeffery RW, Wing RR, Sherwood NE, Tate DF. Physical activity and weight loss: does prescribing higher physical activity goals improve outcome? Am J Clin Nutr. 2003 Oct;78(4):684-9. doi: 10.1093/ajcn/78.4.684. PMID 14522725
- [Background] Wing RR, Jeffery RW. Prescribed "breaks" as a means to disrupt weight control efforts. Obes Res. 2003 Feb;11(2):287-91. doi: 10.1038/oby.2003.43. PMID 12582226
- [Background] Raynor HA, Polley BA, Wing RR, Jeffery RW. Is dietary fat intake related to liking or household availability of high- and low-fat foods? Obes Res. 2004 May;12(5):816-23. doi: 10.1038/oby.2004.98. PMID 15166302
- [Background] Raynor HA, Jeffery RW, Tate DF, Wing RR. Relationship between changes in food group variety, dietary intake, and weight during obesity treatment. Int J Obes Relat Metab Disord. 2004 Jun;28(6):813-20. doi: 10.1038/sj.ijo.0802612. PMID 15037882